CLINICAL TRIAL: NCT00003009
Title: A Phase I Study of Inhalation of Interleukin-2 (IL-2) in Patients With Metastatic or Unresectable Cancer
Brief Title: Inhaled Interleukin-2 in Treating Patients With Metastatic or Unresectable Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065584 (0I-95-1); LAC-USC-0I951; NCI-G97-1264
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Giving interleukin-2 in different ways may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of inhaled interleukin-2 in treating patients with metastatic or unresectable cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the safe and tolerance of an inhaled interleukin-2 (IL-2) administered once or twice a day. II. Determine blood levels of IL-2 and whether there is detectable stimulation of immune cells in patients receiving inhalation IL-2. III. Determine whether there is any shrinkage of pulmonary lesions of patients treated on this study.

OUTLINE: This is a two arm, escalating dose study of interleukin-2 (IL-2). In Arm I patients in cohorts of 3-6 are administered daily inhalations of IL-2 over 15 minutes on Monday through Friday for 4 consecutive weeks. At least 3 patients are treated at each dose level, and all patients in a cohort are observed for at least 2 weeks before escalating to a higher dose in absence of dose limiting toxicity. Escalation stops when maximum tolerated dose (MTD) is determined. In Arm II the initial dose is 25 percent of the MTD determined in Arm I administered by inhalation twice daily on Monday through Friday for 4 weeks. Subsequent patient cohorts receive doses escalated by 33 percent above the previous dose level. Responding patients continue treatment cycles of 4 weeks with 2 weeks of rest until they develop progressive disease or intolerable toxicity. Stable patients may stay on treatment for a maximum of 4 cycles.

PROJECTED ACCRUAL: A minimum of 12-15 and a maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable or metastatic cancer Confirmed by biopsy or fine needle aspiration Tumors must predominantly involve the lung Measurable or evaluable disease No lymphomas or leukemias No AIDS associate Kaposi's Sarcoma No uncontrolled brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-1 Life expectancy: At least 3 months Hematopoietic: WBC at least 4,000/mm3 Platelet count within normal limits Hepatic: Bilirubin no greater than 2 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: Adequate cardiovascular system with NYHA Class 0 or I No uncontrolled cardiac arrhythmias Pulmonary: FEV1 at least 65% of predicted FVC at least 65% of predicted No asthma or bronchial obstruction that would prevent the delivery of IL-2 to all lobes of the lung Other: HIV negative No medical or psychological criteria that would make patient unable to tolerate the treatment Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior interleukin-2 Prior biologic response therapy allowed No chronic use of immunosuppressive medicines Chemotherapy: Prior chemotherapy allowed Endocrine therapy: No chronic steroid use Prior hormonal therapy allowed Radiotherapy: No prior or concurrent radiotherapy except as palliative to areas of painful metastases outside the lung Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1996-02; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond A. Kempf, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States